CLINICAL TRIAL: NCT00676507
Title: Phase III Study of Lucanix™ (Belagenpumatucel-L) in Advanced Non-small Cell Lung Cancer: An International Multicenter, Randomized, Double-blinded, Placebo-controlled Study of Lucanix™ Maintenance Therapy for Stages III/IV NSCLC Subjects Who Have Responded to or Have Stable Disease Following One Regimen of Front-line, Platinum-based Combination Chemotherapy
Brief Title: Phase III Lucanix™ Vaccine Therapy in Advanced Non-small Cell Lung Cancer (NSCLC) Following Front-line Chemotherapy
Acronym: STOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovaRx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NR001-03; BB-IND 8868; NCT00641966 (obsolete NCT alias)
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Lung Neoplasm; Carcinoma Non-small Cell Lung Cancer Stage IIIA; Carcinoma Non-small Cell Lung Cancer Stage IIIB; Carcinoma Non-small Cell Lung Cancer Stage IV
Keywords: Gene therapy; Flow cytometry; Immunoenzyme technique; Laboratory biomarker analysis; Quality-of-life-assessment; Tumor cell-derivative vaccine therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — belagenpumatucel L

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Treatment Arm: This course of therapy is Best Support Care (BSC) plus monthly intradermal (ID) injections of Lucanix™ (belagenpumatucel-L) consisting of 25,000,000 cells in a volume of 0.40 mL.
  Interventions: Biological: Lucanix™
- Control Arm (Placebo Comparator): Control Arm: This course of therapy is Best Support Care (BSC) plus a placebo injection that consists of 0.15% Intralipid® in solution composed of the cryopreservation formulation minus the gene modified cells and dimethyl sulfoxide (DMSO) in a volume of 0.40 mL.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: Lucanix™ — Treatment Arm: Subjects receive Lucanix™ (belagenpumatucel-L) intradermally (ID) once monthly for 18 months and then once at 21 and 24 months in the absence of disease progression or unacceptable toxicity.
  Other Names: belagenpumatucel-L
  Arms: Treatment
Other: Placebo Comparator — Control Arm: Subjects receive placebo ID once monthly for 18 months and then once at 21 and 24 months in the absence of disease progression or unacceptable toxicity.
  Arms: Control Arm

SUMMARY:
Rationale: Vaccines made from gene-modified tumor cells may help the body build an immune response to kill tumor cells. It is not yet known whether vaccine therapy is more effective than a placebo as maintenance therapy in treatment of subjects with non-small cell lung cancer.

Purpose: This randomized phase III trial is studying vaccine therapy to see how well it works compared with a placebo in treating subjects with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
Primary Efficacy Endpoints:

* Compare the overall survival of subjects with stage III or IV non-small cell lung cancer treated with belagenpumatucel-L (Lucanix™) vs placebo.

Secondary Efficacy Endpoints:

* Evaluate the progression free survival (PFS) of subjects treated with Lucanix™ compared to treatment within the BSC control group.
* Evaluate the quality of life (QOL) as determined by the Lung Cancer Symptom Scale (LCSS) compared to treatment within the BSC control group.
* Evaluate the time-to-progression of subjects treated with Lucanix™ compared to treatment within the BSC control group.
* Evaluate the best overall tumor response in subjects treated with Lucanix™ compared to treatment in the BSC control group.
* Evaluate the response duration in subjects treated with Lucanix™ compared to the BSC control group.
* Evaluate the rate of CNS metastases development in subjects treated with Lucanix™ as compared to the BSC control group.
* Adverse events of subjects treated with Lucanix™ will be compared to subjects in the control group.

Outline: This is a multicenter study. Subjects are stratified according to disease stage (IIIA vs IIIB or IV), response to prior treatment with front-line chemotherapy (stable disease vs partial response or complete response), prior treatment with front-line chemotherapy and radiotherapy (front-line chemotherapy with radiotherapy vs front-line chemotherapy alone), and prior treatment with front-line chemotherapy and other anticancer therapy (front-line chemotherapy with bevacizumab vs front-line chemotherapy alone or in combination with another anticancer agent). Subjects are randomized to 1 of 2 treatment arms.

* Treatment Arm: Subjects receive belagenpumatucel-L (Lucanix™) intradermally (ID) once monthly for 18 months and then once at 21 and 24 months in the absence of disease progression or unacceptable toxicity.
* Control Arm: Subjects receive placebo ID once monthly for 18 months and then once at 21 and 24 months in the absence of disease progression or unacceptable toxicity.

Blood samples are collected and analyzed for routine chemistry, cytokines, chemokines, and some instances circulating tumor cells, including response to multiple lung cancer-associated antigens by IFN-γ ELISPOT CD8+ assay; CEA by CD4 class II assay; lung tumor-associated antigens by in vitro proliferation assays; regulatory T-cell (Treg) phenotype by flow cytometry; and Treg function.

Subjects complete the Lung Cancer Symptom Scale quality of life questionnaire at baseline, on the days of treatment, 30 days after completion of study treatment, and then every 3 months for 1 year.

After completion of study treatment, subjects are followed every 3 months for 1 year and then annually for 4 years.

In two phase II trials, many subjects who received Lucanix™ at the same dose that will be administered in this trial had long-term disease stability with a good quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed NSCLC who meet one of the following staging requirements:
* Stage IIIA (T3N2 only) or
* Stage IIIB or
* Stage IV.
* Subjects must have stable disease (SD) or an objective response (PR or CR) to a prior single, frontline, platinum-based chemotherapy regimen (additional prior adjuvant chemotherapy is permitted) consisting of up to six (6) treatment cycles with or without concomitant radiation therapy.
* Not less than four weeks nor more than four months must have elapsed since the completion of the last chemotherapy cycle and registration into the study.
* Subjects treated for brain metastasis(es) are eligible if they have been stable for ≥ 2 months.
* Signed informed consent.
* Not less than 18 years and not more than 75 years old.
* Estimated life expectancy of at least 12 weeks.
* Performance status (ECOG) ≤ 2.
* Absolute neutrophil count ≥ 1,500/mm3.
* Hemoglobin ≥ 9 g/dL.
* Platelet count ≥ 100,000/mm3.
* Albumin levels ≥ 2.5 g/dL.
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN).
* Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 1.5 × ULN.
* Creatinine ≤ 1.5 × ULN.
* Alkaline phosphatase ≤ 5 × ULN.

Exclusion Criteria:

* Concurrent systemic steroids > 2 mg /day prednisone (or prednisone-equivalent of prednisolone or dexamethasone).
* Prior splenectomy.
* Any surgery involving general anesthesia < 4 weeks prior to study registration.
* Chemotherapy more than 4 months or less than 4 weeks prior to study registration.
* Steroid therapy (excluding ≤ 2 mg/day prednisone or prednisone-equivalent of prednisolone or dexamethasone), radiation therapy, or immunotherapy less than 4 weeks prior to study registration.
* Subjects with documented active brain metastasis(es) at the time of study entry are ineligible. However, subjects treated for brain metastasis(es) are eligible if they have been stable for ≥ 2 months.
* Painful bone metastases, or bone metastases that require immediate therapy.
* Significant and/or symptomatic pleural effusions. Presence of clinically detectable (by physical exam) third-space fluid collections, for example, pleural effusions that cannot be controlled by previous chemotherapy and/or drainage, or other procedures, prior to study entry.
* Known allergies to eggs or soy.
* Significant weight loss (≥ 10% body weight in preceding 6 weeks).
* Known HIV positivity (EBV origin of replication in the pCHEK/HBA2 vector used to modify the vaccine components can trans-activate HIV).
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections) or other conditions that, in the opinion of the investigator, would compromise study objectives.
* NCI CTC Grade 3 or 4 peripheral neuropathy at study registration.
* Prior other malignancies (excluding non-melanoma carcinomas of the skin) unless in remission for ≥ 2 years.
* History of psychiatric disorder that would impede ability to give informed consent or adherence to study requirements.
* Pregnant or nursing women, or refusal to practice contraception if of reproductive potential.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Known active Epstein-Barr infection within ≤ 60 days of study registration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2008-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Compare the overall survival of subjects with stage III or IV non-small cell lung cancer treated with belagenpumatucel-L (Lucanix™) vs placebo. | 7 years

SECONDARY OUTCOMES:
Evaluate the progression free survival (PFS) of subjects treated with Lucanix™ compared to treatment within the Best Support Care control group. | 3 years
Evaluate the quality of life (QOL) as determined by the Lung Cancer Symptom Scale (LCSS) compared to treatment within the Best Supportive Care control group. | 3 years
Evaluate the time-to-progression of subjects treated with Lucanix™ compared to treatment within the Best Supportive Care control group. | 3 years
Evaluate the best overall tumor response in subjects treated with Lucanix™ compared to treatment in the Best Supportive Care control group. | 3 years
Evaluate the response duration in subjects treated with Lucanix™ compared to the Best Supportive Care control group. | 3 years
Evaluate the rate of CNS metastases development in subjects treated with Lucanix™ as compared to the Best Supportive Care control group. | 7 years
Adverse events of subjects treated with Lucanix™ will be compared to subjects in the Best Supportive Care control group. | 7 years

CONTACTS AND LOCATIONS:
Locations (80):
- United States (51):
  - Southern Cancer Center, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - Clopton Clinic Hematology/Oncology, Jonesboro, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - University of California, San Diego, La Jolla, California
  - UCLA Pasadena Oncology, Pasadena, California
  - Cancer Care Associates, Redondo, California
  - Innovative Research Center of California, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Cancer Center, Santa Monica, California
  - UCLA Cancer Center-Valencia, Valencia, California
  - UCLA Cancer Center, Westlake Village, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - Pasco Hernando Oncology Associates, P.A., Brooksville, Florida
  - Medical Specialist of Palm Beaches, Lake Worth, Florida
  - Ocala Oncology, Ocala, Florida
  - Space Coast Medical Center, Titusville, Florida
  - Atlanta Cancer Care, Roswell, Georgia
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - St. Francis Medical Group Oncology and Hematology Specialists, Indianapolis, Indiana
  - Iowa Blood and Cancer Center, Cedar Rapids, Iowa
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - National Cancer Institute Center for Cancer Research, Medical Oncology Branch, Bethesda, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Tennessee Cancer Institute, Southaven, Mississippi
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Richmond University Medical Center, Staten Island, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Allergy Partners of West North Carolina, Asheville, North Carolina
  - Cancer Care of WNC, Asheville, North Carolina
  - Gabrail Cancer Center Research LLC, Canton, Ohio
  - Optim Oncology, Midwest City, Oklahoma
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - University of Tennessee Cancer Institute, Bartlett, Tennessee
  - University of Tennessee Cancer Institute, Germantown, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Texas Cancer Center Abilene, Texas Oncology P.A., Abilene, Texas
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Allison Cancer Center, Texas Oncology, P.A., Midland, Texas
  - Tyler Cancer Center, Texas Oncology, Tyler, Texas
  - Seattle Cancer Care Alliance/Fred Hutchinson Cancer Res Ctr/Univ. of Washington Med Ctr, Seattle, Washington
  - Davis Memorial Cancer Care Center, Elkins, West Virginia
  - Marshfield Clinic Weston Center, Weston, Wisconsin
- Canada (2):
  - University of Alberta Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
- Hungary (7):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Semmelweis Egyetem Pulmonológiai Klinika, Budapest
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkórháza, Deszk
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Oktató Kórháza, Nyíregyháza
  - Fejér Megyei Szent György Kórház, Székesfehérvár
  - Pest Megyei Tüdőgyógyintézet, Törökbálint
- India (4):
  - Gujarat Cancer Hospital and Research Institute, Ahmedabad
  - SEAROC Cancer Center, S.K., Jaipur
  - Tata Memorial Hospital, Mumbai
  - Noble Hospital, Pune
- Netherlands (4):
  - Ziekenhuis Groep Twente - locatie Twenteborg Ziekenhuis, Almelo
  - Academisch Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Universitair Medisch Centrum Maastricht, Maastricht
- Poland (5):
  - Akademickie Centrum Kliniczne Szpital Akademii Medycznej w Gdansku, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Wielkopolskie Centrum Pulmunologii i Torakochirurgii, Poznan
  - Centrum Onkologii - Instytut im.Marii Sklodowskiej-Curie, Warsaw
  - Dolnoslaskie Centrum Chorob Pluc, Wroclaw
- Serbia (3):
  - Klinicko-bolnicki centar Bezanijska kosa, Belgrade
  - Institute for pulmonary disease Sremska Kamenica, Kamenitz
  - Klinicki Centar Nis, Niš
- United Kingdom (4):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Glasgow
  - Clatterbridge Centre for Oncology, Bebington, Wirral
  - Ninewells Hospital and Medical School, Dundee
  - Guy's Hospital, London

REFERENCES:
- [Background] Fakhrai H, Mantil JC, Liu L, Nicholson GL, Murphy-Satter CS, Ruppert J, Shawler DL. Phase I clinical trial of a TGF-beta antisense-modified tumor cell vaccine in patients with advanced glioma. Cancer Gene Ther. 2006 Dec;13(12):1052-60. doi: 10.1038/sj.cgt.7700975. Epub 2006 Jul 7. PMID 16826191
- [Background] Nemunaitis J, Nemunaitis M, Senzer N, Snitz P, Bedell C, Kumar P, Pappen B, Maples PB, Shawler D, Fakhrai H. Phase II trial of Belagenpumatucel-L, a TGF-beta2 antisense gene modified allogeneic tumor vaccine in advanced non small cell lung cancer (NSCLC) patients. Cancer Gene Ther. 2009 Aug;16(8):620-4. doi: 10.1038/cgt.2009.15. Epub 2009 Mar 13. PMID 19287371
- [Result] Nemunaitis J, Dillman RO, Schwarzenberger PO, Senzer N, Cunningham C, Cutler J, Tong A, Kumar P, Pappen B, Hamilton C, DeVol E, Maples PB, Liu L, Chamberlin T, Shawler DL, Fakhrai H. Phase II study of belagenpumatucel-L, a transforming growth factor beta-2 antisense gene-modified allogeneic tumor cell vaccine in non-small-cell lung cancer. J Clin Oncol. 2006 Oct 10;24(29):4721-30. doi: 10.1200/JCO.2005.05.5335. Epub 2006 Sep 11. PMID 16966690
- [Derived] Giaccone G, Bazhenova LA, Nemunaitis J, Tan M, Juhasz E, Ramlau R, van den Heuvel MM, Lal R, Kloecker GH, Eaton KD, Chu Q, Dunlop DJ, Jain M, Garon EB, Davis CS, Carrier E, Moses SC, Shawler DL, Fakhrai H. A phase III study of belagenpumatucel-L, an allogeneic tumour cell vaccine, as maintenance therapy for non-small cell lung cancer. Eur J Cancer. 2015 Nov;51(16):2321-9. doi: 10.1016/j.ejca.2015.07.035. Epub 2015 Aug 14. PMID 26283035
- See also: Main sponsor website — http://www.novarx.com
- See also: Clinical trial information — http://www.novarx.com/clinical-trials.php